CLINICAL TRIAL: NCT04203771
Title: Effect of Probiotic Intervention With Lactobacillus Brevis KABP052 (CECT7480) and Lactobacillus Plantarum KABP051 (CECT7481) After Surgical Removal of Mandibular Third Molars: a Randomized, Controlled, Double-blinded Trial
Brief Title: Probiotic Intervention After Surgical Removal of Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Hospital de Nens de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-0202015-FHNB
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Surgery--Complications; Molar, Third
Keywords: Probiotic; Molar removal surgery; Oral pain; Maxillofacial surgery
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Probiotic and placebo tablets with identical appearance were provided in anonymous packages to the investigators, solely labelled with the volunteer's randomization number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Orodispersible tablets containing AB-DENTALAC probiotic formula.
  Interventions: Dietary Supplement: Probiotic AB-DENTALAC; Procedure: Surgical removal of mandibular third molars at baseline; Drug: Ibuprofen
- Control (Placebo Comparator): Orodispersible tablets without probiotic strains (excipients only).
  Interventions: Other: Placebo; Procedure: Surgical removal of mandibular third molars at baseline; Drug: Ibuprofen

INTERVENTIONS:
Dietary Supplement: Probiotic AB-DENTALAC — Orodispersible tablets containing Lactobacillus plantarum [now Lactoplantibacillus plantarum] KABP051 (CECT7481) and Lactobacillus brevis [now Levilactobacillus brevis] KABP052 (CECT7480) as active ingredients, at a minimum dose of 5x10^8 cfu each, and sorbitol (E420) and guar gum (E412) as excipients, taken b.i.d. for 7 days.
  Arms: Probiotic
Other: Placebo — Orodispersible tablets made of sorbitol (E420) and guar gum (E412), taken b.i.d for 7 days.
  Arms: Control
Procedure: Surgical removal of mandibular third molars at baseline — Surgical removal of both mandibular third molars, performed under intravenous sedation and loco-regional anesthesia (Articaine Hydrochloride 4% with Epinephrine 1:100.000), after having undergone a professional oral cleaning.
Drug: Ibuprofen — Ibuprofen syrup at 20-30 mg/Kg of body weight, orally every 8 hours (t.i.d), for 7 days
  Other Names: Dalsy

SUMMARY:
Single-center, double-blind, randomized trial of probiotics L. plantarum KABP-051 (CECT7481) and L. brevis KABP-052 (CECT7480) taken twice daily for 7 days after surgical removal of both mandibular 3rd molars. Patients were assessed for surgery-derived complications in a follow-up visit 7 days after surgery, and provided daily evaluations of pain, swelling and eating difficulty in a patient diary.

DETAILED DESCRIPTION:
This was a single-centre, prospective, double-blind, randomized, placebo-controlled, parallel-group study to evaluate whether probiotic supplementation during 1 week after surgery reduced post-surgery complications compared to placebo.

Healthy subjects of both genders aged between 14 and 25 years who required the surgical removal of both mandibular 3rd molars were recruited from the department of Oral and Maxillofacial Surgery at the Foundation of Hospital de Nens de Barcelona (Children's Hospital of Barcelona).

Patients were randomly assigned to receive probiotic tablets containing a mixture of L. plantarum KABP-051 (CECT7481) and L. brevis KABP-052 (CECT7480) or to receive placebo, twice a day for 7 days post surgery.

Patients were assessed by trained specialists for surgery-derived complications (fever, oral alveolitis, alveolar osteitis, trismus) in a follow-up visit 7 days after surgery. Patients also provided daily evaluations for pain, swelling and eating difficulties in a patient diary.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male and female undergoing surgical removal of both third mandibular molars.
* Aged between 14 and 25 years.
* Providing informed consent if 18yr and older, or parents/guardians providing informed consent otherwise

Exclusion Criteria:

* Subjects with gingival index (GI; according to Loe and Silness. 1963) or dental plaque index (PlI; according to Silness and Loe. 1964) above 2 in the CPI Community Periodontal Index) teeth subset.
* Subjects having used probiotics or antibiotics within 30 days prior to study enrollment.
* Tobacco use
* Pregnant and breastfeeding women.
* Known allergies to ingredients in study products.
* Not willing to refrain from using mouthwashes during the study period

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Complications derived from surgical removal of both mandibular third molars | 7 days
  Occurrence of low grade fever (Yes/No), oral alveolitis (Yes/No) and/or trismus (Yes/No), as determined by a trained specialist

SECONDARY OUTCOMES:
Post-surgical pain, patient-rated | Daily, for 7 days
  Oral pain derived from surgery, rated 0 (none) to 10 (unbearable) in a Visual Analog Scale (VAS) in a patient diary.
Post-surgical swelling, patient-rated | Daily, for 7 days
  Mandibular swelling derived from surgery, rated 0 (none) to 10 (unbearable) in a Visual Analog Scale (VAS) in a patient diary.
Post-surgical eating difficulty, patient-rated | Daily, for 7 days
  Eating difficulty as a result from surgery, rated 0 (none) to 10 (unbearable) in a Visual Analog Scale (VAS) in a patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Ferres Padro, MD, Principal Investigator — Children's Hospital of Barcelona; Jordi Espadaler Mazo, PhD, Study Chair — AB Biotics, SA
Locations (1):
- Hospital de Nens de Barcelona (Children's Hospital of Barcelona)), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No